CLINICAL TRIAL: NCT05690178
Title: Effect of Deep Tissue Massage on Subjective and Objective Parameters in Office Workers With Chronic Low Back Pain
Brief Title: Deep Tissue Massage in Office Workers With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Principal Investigator, Michał Wendt, Principal Investigator, Poznan University of Physical Education
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DTM-CLBP-OW
Record Dates: First submitted 2023-01-01; First posted 2023-01-19 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Chronic Low-back Pain
Keywords: Chronic Low-back Pain; Range of motion; Pressure pain threshold; Myoton; Muscle properties; Surface electromyography; Oswestry Disability Index; Rolland Morris Disability Questionnaire; Disability; Visual Analogue Scale; Deep Tissue Massage; Manual Therapy

STUDY DESIGN:
Intervention Model Description: The first step was recruitment. Based on the qualifying and disqualifying criteria, 40 people were selected. Each participant was randomly assigned to a specific group (Deep Tissue Massage (DTM) experimental group or control group). Initial measurements were collected from all participants. Participants in the DTM group had therapy, while those in the control group had no therapy. The therapist was responsible for performing the DTM therapy. Each participant in the experimental group received 4 treatments (45 minutes each, 3 days between them) over a period of 2 weeks. After the end of the whole therapy, final measurements were made. The researcher was responsible for taking measurements for each participant. The person acting as the coordinator supervised the proper course of the research. The collected data was analyzed by a person evaluating the results.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (participant, researcher, outcome assessor). Participants did not know which study group they belonged to. Each participant drew a number that was characteristic of a given research group (experimental DTM group or control group). The researcher also did not know which group the participant belonged to (he only used the participant number). Outcome assessor did not know which group was experimental and which was control (they were marked with numbers instead of names). The coordinator supervised the proper course of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DTM group (Experimental): This group of participants (N=20) received Deep Tissue Massage therapy.
  Interventions: Other: Deep Tissue Massage
- Control group (No Intervention): This group of participants (N=20) did not receive any intervention.

INTERVENTIONS:
Other: Deep Tissue Massage — The Deep Tissue Massage lasted 45 minutes. The entire therapy included 4 treatments over a period of 2 weeks. The interval between treatments was 3 days. The conducted therapy included techniques for: quadratus lumborum muscle, erector spinae muscle, thoracolumbar fascia, iliopsoas muscle. All techniques were performed on both sides of the patient's body.
  Arms: DTM group

SUMMARY:
The main objective of the study was to assess the impact of deep tissue massage on subjective and objective parameters in a group of office workers with chronic low back pain.

Specific objectives:

* Assessment of the impact of deep tissue massage on the level of pain
* Assessment of the impact of deep tissue massage on the level of disability
* Assessment of the impact of deep tissue massage on the mobility of the lumbar spine
* Assessment of the effect of deep tissue massage on the discomfort threshold of tissue compression in the area of the erector spinae muscle
* Assessment of the impact of deep tissue massage on the biophysical parameters of the soft tissues of the erector spinae muscle
* Evaluation of the impact of deep tissue massage on the bioelectric potentials of the erector spinae muscle during everyday activities and the flexion-relaxation test

Hypotheses:

* Deep tissue massage will reduce the level of pain in the lumbar spine
* Deep tissue massage will reduce the level of disability
* Deep tissue massage will increase the range of motion of the lumbar spine in all directions
* Deep tissue massage will reduce the threshold of discomfort when compressing the soft tissues of the erector spinae muscle
* Deep tissue massage will reduce muscle tone and stiffness and increase the elasticity of the back extensor muscle
* Deep tissue massage will increase the bioelectrical potentials of the erector spinae muscle while performing tests of activities of daily living
* Deep tissue massage will reduce the value of the flexion-relaxation test

DETAILED DESCRIPTION:
Deep tissue massage is a manual action of the therapist in the superficial and deep layers of muscles and fascia in order to relax, change abnormal patterns, eliminate tension and pain in a maximally ergonomic way. Deep tissue massage should be described as an independent method of therapy using a specific set of techniques and principles. It is a safe method with a wide range of applications, while the techniques themselves can be modified to the needs of the patient. It is believed that deep tissue massage causes: improvement of tissue blood supply, reduction of muscle tension, stretching of muscles and fascia, improvement of muscle and joint function.

Participants A total of 40 patients (30 to 60 years of age) participated in the study. All participants were characterized by the presence of chronic low back pain syndrome, performed office work for 8 hours a day and were characterized by moderate physical activity. Using randomization, participants were divided into two groups (experimental and control). The experimental group included participants who received deep tissue massage (N=20, 18 women and 2 men, average age: 40). The control group included participants who did not receive therapy (N=20, 13 women and 7 men, average age: 43).

Intervention The deep tissue massage lasted 45 minutes. The entire therapy included 4 treatments over a period of 2 weeks. The interval between treatments was 3 days. The conducted therapy included techniques for: quadratus lumborum muscle, erector spinae muscle, thoracolumbar fascia, iliopsoas muscle. All techniques were performed on both sides of the patient's body.

Research methods

The following measurement equipment was used to collect the data:

1. Electrogoniometer. Penny & Giles strain gauge electrogoniometer with two sensors (SG150 - two-axis, Q110 - single-axis). Measurements were taken in a standing position, in accordance with the measurement methodology according to Lewandowsky. All movements of the lumbar spine (forward bending, backward bending, right bending, left bending, right rotation, left rotation) were examined. The average of the three measurements was the result of movability for a given direction. The sensors were attached to the skin using Biometrics double-sided tape. The upper sensor was placed on the Th12 spinous process (lower edge of the sensor), while the lower sensor was mounted on the base of the sacrum (upper edge).
2. Algometer. The Wagner Instruments algometer was used to assess the subjective parameter, i.e. the first discomfort threshold. In the study, the measurement site was the point located on the longissimus muscle, which is a component of the erector spinae muscle. The subjects lay in front. The pressure, detected by the algometer sensor, was applied from above and perpendicularly to the examined muscle (two fingers laterally from the L1 spinous process). Three measurements were made alternately for both sides of the examined muscle. From these measurements, mean values were calculated, which were the results for the right and left sides of the examined muscle.
3. MyotonPRO. In order to study the biophysical parameters of soft tissues, i.e. muscle tone (F) [Hz], stiffness (S) [N/m] and elasticity (D) [no units], the MyotonPRO apparatus was used. During the measurements, the tested person lay on his front. Measurements were made on the longissimus muscle (2 fingers lateral to the L1 spinous process). The pattern composer was programmed as follows: tapping time: 15 ms, interval: 0.8 s, mode: multiscan (5 repetitions). Measurements were made on the right and left muscles.
4. Kinesiologic electromyography (EMG). Kinesiologic electromyography was carried out with an 8-channel electromyographic system with plate electrodes (model W4X8, Biometrics Ltd). The results were recorded using DataLog Bluetooth V7.5 software (Biometrics Ltd). During the examination, six multiple-use surface electrodes (type SX230 1000) were attached with an adhesive tape, after removal of body hair froma 2 cm x 1 cm area of intact skin, disinfection of electrode surface, and wiping the skin a few times with salicylic alcohol to reduce its resistance. The reference electrode (type R230, Biometrics Ltd) was fixed at the distal end of the radius (Lister's tubercle region) with an elastic band. The examination involved lumbar segment of the longissimus muscle, iliocostalis and multifidus (both right- and left-sided bundles). The electrodes were placed according to the international guidelines published by SENIAM. The examination was painless and noninvasive and did not require subject's exposure to any additional electric stimulation. The measurement was preceded by a 10-min warm-up of the keymuscle groups. The list of determined electromyographic parameters included the amplitude of bioelectrical signal from the longissimus, iliocostalis and multifidus muscles, expressed in microvolt. Avoiding a confounding effect associated with measurement conditions, the results were normalized to a reference Maximum Voluntary Contraction (MVC) and expressed in percent. After fixation of the electrodes and preparation of the system, MVC of the longissimus, iliocostalis and multifidus were determined according to the international SENIAM guidelines. The examination started with the subject lying down in a prone position, with arms crossed under the chin, and extended legs. The EMG recordings were obtained during three active extensions of the spine, each lasting 3 seconds, with 30-second intervals in between. MVCs , corresponding to 100% neuromuscular activation of the muscles, was calculated as the mean amplitude for the three repetitions (for each muscle). At the beginning, the Flexion-Relaxation (FR) test was performed. The participant performed forward flexion of the spine and hung freely in this position for 10 seconds. During this test, the participant was asked to be as relaxed as possible. Then the participant was tested during successive tests of activities of daily living: getting up from a chair, sitting on it, lifting and lowering a 1 kg and 2 kg weight. Each test was run at an individually adjusted pace and consisted of three repetitions with 30-second rests between them. The test started at the investigator's request. While lifting and lowering the weights, the subjects kept a straight back, and each hold of the weight lasted 3 seconds and was performed on straight elbows. The result of each test is presented as the mean amplitude for three repetitions for each muscle. The results were normalized to the MVC to assess the degree of muscle involvement during various activities (standing up, sitting down, raising and lowering the roller) in relation to maximal neuromuscular activation. To ensure accurate results, the correct attachment of each electrode was rechecked before each repetition.
5. Revised Oswestry Pain Questionnaire (ODI). The degree of LBP imposed limitations in activity of daily ling (ADLs) was determined with Revised Oswestry Pain Questionnaire, also referred to as Oswestry Disability Index (ODI). The survey consisted of 10 questions, each with 6 possible responses scored from 0 to 5 points. If the respondent chose more than one answer to a given question, the one with higher score was recorded and subjected to the analysis. Maximum overall score amounted to 50 points, which corresponded to 100% disability due to lumbar pain.
6. Roland-Morris Disability Questionnaire (RMDQ). The instrument consists of 24 statements about pain and its influence on ADLs. The respondent chooses only the statements that refer to his/her ailments. Maximum overall score may vary between 0 and 24 points.
7. Visual-Analog Scale (VAS). This subjective tool is used to assess the level of pain. The participant marks the level of pain on a 10 cm scale, where 0 is no pain and 10 is the maximum pain he has ever felt.

In order to assess the impact of deep tissue massage therapy on the study population, two measurements were made over time: before and after therapy.

Ethics All measurement methods used were non-invasive and safe for health. The study was approved by the local Bioethics Committee. Each participant had the right to withdraw from the study at any stage. All collected data is anonymous and will be used only to conduct statistical analyzes for scientific purposes.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Low-Back Pain
* office worker

Exclusion Criteria:

* spine surgeries
* cauda equina syndrome
* cancer
* pain or motor and sensory deficits in the lower extremities below the level of the knee
* various therapies to treat chronic low-back pain

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Lumbar anterior flexion (PRE) | Through study completion, an average of 2 weeks.
  Electrogoniometric measurement of the angular range of motion the day before the therapy
Lumbar anterior flexion (POST) | Through study completion, an average of 2 weeks.
  Electrogoniometric measurement of the angular range of motion the day after the therapy
Lumbar posterior flexion (PRE) | Through study completion, an average of 2 weeks.
  Electrogoniometric measurement of the angular range of motion the day before the therapy
Lumbar posterior flexion (POST) | Through study completion, an average of 2 weeks.
  Electrogoniometric measurement of the angular range of motion the day after the therapy
Lumbar right flexion (PRE) | Through study completion, an average of 2 weeks.
  Electrogoniometric measurement of the angular range of motion the day before the therapy
Lumbar right flexion (POST) | Through study completion, an average of 2 weeks.
  Electrogoniometric measurement of the angular range of motion the day after the therapy
Lumbar left flexion (PRE) | Through study completion, an average of 2 weeks.
  Electrogoniometric measurement of the angular range of motion the day before the therapy
Lumbar left flexion (POST) | Through study completion, an average of 2 weeks.
  Electrogoniometric measurement of the angular range of motion the day after the therapy
Lumbar right rotation (PRE) | Through study completion, an average of 2 weeks.
  Electrogoniometric measurement of the angular range of motion the day before the therapy
Lumbar right rotation (POST) | Through study completion, an average of 2 weeks.
  Electrogoniometric measurement of the angular range of motion the day after the therapy
Lumbar left rotation (PRE) | Through study completion, an average of 2 weeks.
  Electrogoniometric measurement of the angular range of motion the day before the therapy
Lumbar left rotation (POST) | Through study completion, an average of 2 weeks.
  Electrogoniometric measurement of the angular range of motion the day after the therapy
Stiffness (S) of the right longissimus muscle (PRE) | Through study completion, an average of 2 weeks.
  Myotonometer examination of soft tissue properties the day before the intervention
Stiffness (S) of the right longissimus muscle (POST) | Through study completion, an average of 2 weeks.
  Myotonometer examination of soft tissue properties the day after the therapy
Stiffness (S) of the left longissimus muscle (PRE) | Through study completion, an average of 2 weeks.
  Myotonometer examination of soft tissue properties the day before the therapy
Stiffness (S) of the left longissimus muscle (POST) | Through study completion, an average of 2 weeks.
  Myotonometer examination of soft tissue properties the day after the therapy
Elasticity (D) of the right longissimus muscle (PRE) | Through study completion, an average of 2 weeks.
  Myotonometer examination of soft tissue properties the day before the therapy
Elasticity (D) of the right longissimus muscle (POST) | Through study completion, an average of 2 weeks.
  Myotonometer examination of soft tissue properties the day after the therapy
Elasticity (D) of the left longissimus muscle (PRE) | Through study completion, an average of 2 weeks.
  Myotonometer examination of soft tissue properties the day before the therapy
Elasticity (D) of the left longissimus muscle (POST) | Through study completion, an average of 2 weeks.
  Myotonometer examination of soft tissue properties the day after the therapy
Muscle tone (F) of the right longissimus muscle (PRE) | Through study completion, an average of 2 weeks.
  Myotonometer examination of soft tissue properties the day before the therapy
Muscle tone (F) of the right longissimus muscle (POST) | Through study completion, an average of 2 weeks.
  Myotonometer examination of soft tissue properties the day after the therapy
Muscle tone (F) of the left longissimus muscle (PRE) | Through study completion, an average of 2 weeks.
  Myotonometer examination of soft tissue properties the day before the therapy
Muscle tone (F) of the left longissimus muscle (POST) | Through study completion, an average of 2 weeks.
  Myotonometer examination of soft tissue properties the day after the therapy
Pressure pain threshold (PPT) of the right longissimus muscle (PRE) | Through study completion, an average of 2 weeks.
  Examination of the first discomfort threshold using an algometer the day before the therapy
Pressure pain threshold (PPT) of the right longissimus muscle (POST) | Through study completion, an average of 2 weeks.
  Examination of the first discomfort threshold using an algometer the day after the therapy
Pressure pain threshold (PPT) of the left longissimus muscle (PRE) | Through study completion, an average of 2 weeks.
  Examination of the first discomfort threshold using an algometer the day before the therapy
Pressure pain threshold (PPT) of the left longissimus muscle (POST) | Through study completion, an average of 2 weeks.
  Examination of the first discomfort threshold using an algometer the day after the therapy
EMG - MVC for right longissimus muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of maximal voluntary contraction of the right longissimus muscle the day before therapy
EMG - MVC for right longissimus muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of maximal voluntary contraction of the right longissimus muscle the day after the therapy
EMG - MVC for left longissimus muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of maximal voluntary contraction of the left longissimus muscle the day before the therapy
EMG - MVC for left longissimus muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of maximal voluntary contraction of the left longissimus muscle the day after the therapy
EMG - MVC for right iliocostalis muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of maximal voluntary contraction of the left longissimus muscle the day before the therapy
EMG - MVC for right iliocostalis muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of maximal voluntary contraction of the right iliocostalis muscle the day after the therapy
EMG - MVC for left iliocostalis muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of maximal voluntary contraction of the left longissimus muscle the day before the therapy
EMG - MVC for left iliocostalis muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of maximal voluntary contraction of the left longissimus muscle the day after the therapy
EMG - MVC for right multifidus muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of maximal voluntary contraction of the right multifidus muscle the day before the therapy
EMG - MVC for right multifidus muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of maximal voluntary contraction of the right multifidus muscle the day after the therapy
EMG - MVC for left multifidus muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of maximal voluntary contraction of the left multifidus muscle the day before the therapy
EMG - MVC for left multifidus muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of maximal voluntary contraction of the left multifidus muscle the day after the therapy
EMG - FR test for right longissimus muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the right longissimus muscle during the Flexion-Relaxation test the day before the therapy
EMG - FR test for right longissimus muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the right longissimus muscle during the Flexion-Relaxation test the day after the therapy
EMG - FR test for left longissimus muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left longissimus muscle during the Flexion-Relaxation test the day before the therapy
EMG - FR test for left longissimus muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left longissimus muscle during the Flexion-Relaxation test the day after the therapy
EMG - FR test for right iliocostalis muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left longissimus muscle during the Flexion-Relaxation test the day before the therapy
EMG - FR test for right iliocostalis muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left longissimus muscle during the Flexion-Relaxation test the day after the therapy
EMG - FR test for left iliocostalis muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left longissimus muscle during the Flexion-Relaxation test the day before the therapy
EMG - FR test for left iliocostalis muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left longissimus muscle during the Flexion-Relaxation test the day after the therapy
EMG - FR test for right multifidus muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left longissimus muscle during the Flexion-Relaxation test the day before the therapy
EMG - FR test for right multifidus muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left longissimus muscle during the Flexion-Relaxation test the day after the therapy
EMG - FR test for left multifidus muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left longissimus muscle during the Flexion-Relaxation test the day before the therapy
EMG - FR test for left multifidus muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left multifidus muscle during the Flexion-Relaxation test the day after the therapy
EMG - sitting and standing test for right longissimus muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left multifidus muscle during sitting and standing test the day before the therapy
EMG - sitting and standing test for right longissimus muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the right longissimus muscle during sitting and standing test the day after the therapy
EMG - sitting and standing test for left longissimus muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left longissimus muscle during sitting and standing test the day before the therapy
EMG - sitting and standing test for left longissimus muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left longissimus muscle during sitting and standing test the day after the therapy
EMG - sitting and standing test for right iliocostalis muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the right iliocostalis muscle during sitting and standing test the day before the therapy
EMG - sitting and standing test for right iliocostalis muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the right iliocostalis muscle during sitting and standing test the day after the therapy
EMG - sitting and standing test for left iliocostalis muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left iliocostalis muscle during sitting and standing test the day before the therapy
EMG - sitting and standing test for left iliocostalis muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left iliocostalis muscle during sitting and standing test the day after the therapy
EMG - sitting and standing test for right multifidus muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the right multifidus muscle during sitting and standing test the day before the therapy
EMG - sitting and standing test for right multifidus muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the right multifidus muscle during sitting and standing test the day after the therapy
EMG - sitting and standing test for left multifidus muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left multifidus muscle during sitting and standing test the day before the therapy
EMG - sitting and standing test for left multifidus muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left multifidus muscle during sitting and standing test the day after the therapy
EMG - weight holding test (1 kg) for right longissimus muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the right longissimus muscle during the weight holding test (1kg) the day before the therapy
EMG - weight holding test (1 kg) for right longissimus muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the right longissimus muscle during the weight holding test (1kg) the day after the therapy
EMG - weight holding test (1 kg) for left longissimus muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left longissimus muscle during the weight holding test (1kg) the day before the therapy
EMG - weight holding test (1 kg) for left longissimus muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left longissimus muscle during the weight holding test (1kg) the day after the therapy
EMG - weight holding test (1 kg) for right iliocostalis muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the right iliocostalis muscle during the weight holding test (1kg) the day before the therapy
EMG - weight holding test (1 kg) for right iliocostalis muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the right iliocostalis muscle during the weight holding test (1kg) the day after the therapy
EMG - weight holding test (1 kg) for left iliocostalis muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left iliocostalis muscle during the weight holding test (1kg) the day before the therapy
EMG - weight holding test (1 kg) for left iliocostalis muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left iliocostalis muscle during the weight holding test (1kg) the day after the therapy
EMG - weight holding test (1 kg) for right multifidus muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the right multifidus muscle during the weight holding test (1kg) the day before the therapy
EMG - weight holding test (1 kg) for right multifidus muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the right multifidus muscle during the weight holding test (1kg) the day after the therapy
EMG - weight holding test (1 kg) for left multifidus muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left multifidus muscle during the weight holding test (1kg) the day before the therapy
EMG - weight holding test (1 kg) for left multifidus muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left multifidus muscle during the weight holding test (1kg) the day after the therapy
EMG - weight holding test (2 kg) for right longissimus muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the right longissimus muscle during the weight holding test (1kg) the day before the therapy
EMG - weight holding test (2 kg) for right longissimus muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the right longissimus muscle during the weight holding test (1kg) the day after the therapy
EMG - weight holding test (2 kg) for left longissimus muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left longissimus muscle during the weight holding test (1kg) the day before the therapy
EMG - weight holding test (2 kg) for left longissimus muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left longissimus muscle during the weight holding test (1kg) the day after the therapy
EMG - weight holding test (2 kg) for right iliocostalis muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the right iliocostalis muscle during the weight holding test (1kg) the day before the therapy
EMG - weight holding test (2 kg) for right iliocostalis muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the right iliocostalis muscle during the weight holding test (1kg) the day after the therapy
EMG - weight holding test (2 kg) for left iliocostalis muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left iliocostalis muscle during the weight holding test (1kg) the day before the therapy
EMG - weight holding test (2 kg) for left iliocostalis muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left iliocostalis muscle during the weight holding test (1kg) the day after the therapy
EMG - weight holding test (2 kg) for right multifidus muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the right multifidus muscle during the weight holding test (1kg) the day before the therapy
EMG - weight holding test (2 kg) for right multifidus muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the right multifidus muscle during the weight holding test (1kg) the day after the therapy
EMG - weight holding test (2 kg) for left multifidus muscle (PRE) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left multifidus muscle during the weight holding test (1kg) the day before the therapy
EMG - weight holding test (2 kg) for left multifidus muscle (POST) | Through study completion, an average of 2 weeks.
  Electromyographic measurements of the left multifidus muscle during the weight holding test (1kg) the day after the therapy
Revised Oswestry Pain Questionnaire (PRE) | Through study completion, an average of 2 weeks.
  Revised Oswestry Pain Questionnaire (ODI) - the day before therapy. The minimum score is 0, while the maximum is 50, which proves 100% disability. A higher result is worse and proves the patient's disability in everyday activities.
Revised Oswestry Pain Questionnaire (POST) | Through study completion, an average of 2 weeks.
  Revised Oswestry Pain Questionnaire (ODI) - the day after therapy. The minimum score is 0, while the maximum is 50, which proves 100% disability. A higher result is worse and proves the patient's disability in everyday activities.
Roland-Morris Disability Questionnaire (PRE) | Through study completion, an average of 2 weeks.
  Roland-Morris Disability Questionnaire (RMDQ) - the day before therapy. The minimum score is 0, while the maximum is 24. The higher the score, the worse it is and it illustrates the poor functional condition of the examined person.
Roland-Morris Disability Questionnaire (POST) | Through study completion, an average of 2 weeks.
  Roland-Morris Disability Questionnaire (RMDQ) - the day after therapy. The minimum score is 0, while the maximum is 24. The higher the score, the worse it is and it illustrates the poor functional condition of the examined person.
Visual-Analog Scale (PRE) | Through study completion, an average of 2 weeks.
  Visual-Analog Scale (VAS) - the day before therapy. The minimum score is 0 and the maximum score is 10. The higher the score, the worse it is and it reflects the subjective level of pain experienced.
Visual-Analog Scale (POST) | Through study completion, an average of 2 weeks.
  Visual-Analog Scale (VAS) - the day after therapy. The minimum score is 0 and the maximum score is 10. The higher the score, the worse it is and it reflects the subjective level of pain experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Michał Wendt, PhD, Principal Investigator — Poznan University of Physical Education, Department of Biology and Anatomy
Locations (1):
- Poznan University of Physical Education, Department of Biology and Anatomy, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Yes
University IPD sharing platform is under preparation. All data will also be available to researchers via the principal researcher's email (wendt@awf.poznan.pl) or Research Gate website.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available from May/June 2023.
Access Criteria: Available to all researchers.
URL: https://awf.poznan.pl/uczelnia/wydzialy/wydzial-nauk-o-zdrowiu/katedra-nauk-biologicznych/zaklad-biologii-i-anatomii/pracownicy/

REFERENCES:
- [Background] Willard FH, Vleeming A, Schuenke MD, Danneels L, Schleip R. The thoracolumbar fascia: anatomy, function and clinical considerations. J Anat. 2012 Dec;221(6):507-36. doi: 10.1111/j.1469-7580.2012.01511.x. Epub 2012 May 27. PMID 22630613
- [Background] Williams ACC, Craig KD. Updating the definition of pain. Pain. 2016 Nov;157(11):2420-2423. doi: 10.1097/j.pain.0000000000000613. No abstract available. PMID 27200490
- [Background] Schuenke MD, Vleeming A, Van Hoof T, Willard FH. A description of the lumbar interfascial triangle and its relation with the lateral raphe: anatomical constituents of load transfer through the lateral margin of the thoracolumbar fascia. J Anat. 2012 Dec;221(6):568-76. doi: 10.1111/j.1469-7580.2012.01517.x. Epub 2012 May 15. PMID 22582887
- [Background] Tesarz J, Hoheisel U, Wiedenhofer B, Mense S. Sensory innervation of the thoracolumbar fascia in rats and humans. Neuroscience. 2011 Oct 27;194:302-8. doi: 10.1016/j.neuroscience.2011.07.066. Epub 2011 Aug 2. PMID 21839150
- [Background] Saper RB, Lemaster C, Delitto A, Sherman KJ, Herman PM, Sadikova E, Stevans J, Keosaian JE, Cerrada CJ, Femia AL, Roseen EJ, Gardiner P, Gergen Barnett K, Faulkner C, Weinberg J. Yoga, Physical Therapy, or Education for Chronic Low Back Pain: A Randomized Noninferiority Trial. Ann Intern Med. 2017 Jul 18;167(2):85-94. doi: 10.7326/M16-2579. Epub 2017 Jun 20. PMID 28631003
- [Background] Nakipoglu GF, Karagoz A, Ozgirgin N. The biomechanics of the lumbosacral region in acute and chronic low back pain patients. Pain Physician. 2008 Jul-Aug;11(4):505-11. PMID 18690279
- [Background] Marshall PWM, Schabrun S, Knox MF. Physical activity and the mediating effect of fear, depression, anxiety, and catastrophizing on pain related disability in people with chronic low back pain. PLoS One. 2017 Jul 7;12(7):e0180788. doi: 10.1371/journal.pone.0180788. eCollection 2017. PMID 28686644
- [Background] Maher C, Underwood M, Buchbinder R. Non-specific low back pain. Lancet. 2017 Feb 18;389(10070):736-747. doi: 10.1016/S0140-6736(16)30970-9. Epub 2016 Oct 11. PMID 27745712
- [Background] Le Huec JC, Thompson W, Mohsinaly Y, Barrey C, Faundez A. Sagittal balance of the spine. Eur Spine J. 2019 Sep;28(9):1889-1905. doi: 10.1007/s00586-019-06083-1. Epub 2019 Jul 22. PMID 31332569
- [Background] Koren Y, Kalichman L. Deep tissue massage: What are we talking about? J Bodyw Mov Ther. 2018 Apr;22(2):247-251. doi: 10.1016/j.jbmt.2017.05.006. Epub 2017 May 17. PMID 29861215
- [Background] Cai XY, Sun MS, Huang YP, Liu ZX, Liu CJ, Du CF, Yang Q. Biomechanical Effect of L4 -L5 Intervertebral Disc Degeneration on the Lower Lumbar Spine: A Finite Element Study. Orthop Surg. 2020 Jun;12(3):917-930. doi: 10.1111/os.12703. Epub 2020 May 31. PMID 32476282
- [Background] Bogduk N. On the definitions and physiology of back pain, referred pain, and radicular pain. Pain. 2009 Dec 15;147(1-3):17-9. doi: 10.1016/j.pain.2009.08.020. Epub 2009 Sep 16. No abstract available. PMID 19762151
- [Background] Hansen AE, Marcus NJ. Is It Time to Consider Soft Tissue as a Pain Generator in Nonspecific Low Back Pain? Pain Med. 2016 Nov;17(11):1969-1970. doi: 10.1093/pm/pnw204. Epub 2016 Aug 27. No abstract available. PMID 27570247
- [Result] Zheng Z, Wang J, Gao Q, Hou J, Ma L, Jiang C, Chen G. Therapeutic evaluation of lumbar tender point deep massage for chronic non-specific low back pain. J Tradit Chin Med. 2012 Dec;32(4):534-7. doi: 10.1016/s0254-6272(13)60066-7. PMID 23427384
- [Result] Majchrzycki M, Kocur P, Kotwicki T. Deep tissue massage and nonsteroidal anti-inflammatory drugs for low back pain: a prospective randomized trial. ScientificWorldJournal. 2014 Feb 23;2014:287597. doi: 10.1155/2014/287597. eCollection 2014. PMID 24707200
- [Result] van den Dolder PA, Roberts DL. A trial into the effectiveness of soft tissue massage in the treatment of shoulder pain. Aust J Physiother. 2003;49(3):183-8. doi: 10.1016/s0004-9514(14)60238-5. PMID 12952518
- [Result] van den Dolder PA, Ferreira PH, Refshauge KM. Effectiveness of Soft Tissue Massage for Nonspecific Shoulder Pain: Randomized Controlled Trial. Phys Ther. 2015 Nov;95(11):1467-77. doi: 10.2522/ptj.20140350. Epub 2015 May 28. PMID 26023217
- [Result] Furlan AD, Giraldo M, Baskwill A, Irvin E, Imamura M. Massage for low-back pain. Cochrane Database Syst Rev. 2015 Sep 1;2015(9):CD001929. doi: 10.1002/14651858.CD001929.pub3. PMID 26329399
- [Result] Seffrin CB, Cattano NM, Reed MA, Gardiner-Shires AM. Instrument-Assisted Soft Tissue Mobilization: A Systematic Review and Effect-Size Analysis. J Athl Train. 2019 Jul;54(7):808-821. doi: 10.4085/1062-6050-481-17. Epub 2019 Jul 19. PMID 31322903
- [Result] Best TM, Hunter R, Wilcox A, Haq F. Effectiveness of sports massage for recovery of skeletal muscle from strenuous exercise. Clin J Sport Med. 2008 Sep;18(5):446-60. doi: 10.1097/JSM.0b013e31818837a1. PMID 18806553
- [Result] Bervoets DC, Luijsterburg PA, Alessie JJ, Buijs MJ, Verhagen AP. Massage therapy has short-term benefits for people with common musculoskeletal disorders compared to no treatment: a systematic review. J Physiother. 2015 Jul;61(3):106-16. doi: 10.1016/j.jphys.2015.05.018. Epub 2015 Jun 17. PMID 26093806
- [Result] Kassolik K, Andrzejewski W, Brzozowski M, Wilk I, Gorecka-Midura L, Ostrowska B, Krzyzanowski D, Kurpas D. Comparison of massage based on the tensegrity principle and classic massage in treating chronic shoulder pain. J Manipulative Physiol Ther. 2013 Sep;36(7):418-27. doi: 10.1016/j.jmpt.2013.06.004. Epub 2013 Jul 25. PMID 23891481
- [Result] Romanowski MW, Spiritovic M, Rutkowski R, Dudek A, Samborski W, Straburzynska-Lupa A. Comparison of Deep Tissue Massage and Therapeutic Massage for Lower Back Pain, Disease Activity, and Functional Capacity of Ankylosing Spondylitis Patients: A Randomized Clinical Pilot Study. Evid Based Complement Alternat Med. 2017;2017:9894128. doi: 10.1155/2017/9894128. Epub 2017 Aug 6. PMID 28845185
- [Derived] Wendt M, Rubach J, Waszak M. Short-term effect after soft tissue manipulation session on subjective and objective parameters in office workers with chronic low back pain: A randomized clinical trial. PLoS One. 2025 Nov 21;20(11):e0336685. doi: 10.1371/journal.pone.0336685. eCollection 2025. PMID 41270086
- See also: Recommendations for sensor locations in trunk or (lower) back muscles — http://seniam.org/back_location.htm